CLINICAL TRIAL: NCT03998488
Title: A Randomized, Placebo-controlled Clinical Trial Examining the Efficacy of Fecal Microbiota Transplantation (FMT) and Subsequent Dietary Fiber in Patients With Moderate Ulcerative Colitis
Brief Title: Examining the Efficacy of Fecal Microbiota Transplantation (FMT) and Dietary Fiber in Patients With Ulcerative Colitis
Acronym: MINDFUL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Crohn's and Colitis Foundation (Other); National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 19-04020045; 5R01DK128257 (NIH)
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Results first posted 2024-04-02 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Ulcerative Colitis; Inflammatory Bowel Diseases
Keywords: FMT; Fecal Microbiota Transplantation; Inflammatory Bowel Diseases
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Eligible subjects will be randomly assigned to one of the three (Placebo or Investigational FMT +/- Psyllium) treatment groups. A series of randomized blocks of 6-10 will be generated with a 1:1:1 allocation ratio.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blinded study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Investigational FMT (Experimental): Participants will be blindly randomized to receive a single dose of investigational FMT during the week 0 colonoscopy.
  Additionally, participants will blindly receive a single dose of placebo FMT during the week 8 by flexible sigmoidoscopy.
  Interventions: Drug: Fecal Microbiota Transplantation
- Investigational FMT + psyllium fiber (Active Comparator): Participants will be blindly randomized to receive a single dose of investigational FMT during the week 0 colonoscopy. They will also receive fiber supplementation of 1 teaspoon 2x/day for 8 weeks.
  Additionally, participants will blindly receive a single dose of placebo FMT during the week 8 by flexible sigmoidoscopy.
  Interventions: Drug: Fecal Microbiota Transplantation; Dietary Supplement: Psyllium Husk Powder
- Placebo FMT +/- psyllium fiber (Placebo Comparator): Participants will be blindly randomized to receive a single dose of placebo FMT during the week 0 colonoscopy. They may or may not also receive fiber supplementation of 1 teaspoon 2x/day for 8 weeks.
  Additionally, participants will blindly receive a single dose of investigational FMT during the week 8 by flexible sigmoidoscopy.
  Interventions: Dietary Supplement: Psyllium Husk Powder

INTERVENTIONS:
Drug: Fecal Microbiota Transplantation — The proposed intervention will deliver 250 milliliters of FMT by colonoscopy to the investigational FMT treatment groups at week 0. The placebo treatment group will instead receive the placebo FMT by colonoscopy at week 0 and then the investigational FMT by flexible sigmoidoscopy at week 8.
  Investigational FMT is biologically active human fecal material that is pre-screened, tested, quarantined, stored, packaged, and labeled by OpenBiome. Placebo FMP250 is a control unit made of glycerol, saline, and food dye that is stored, packaged, and labeled identically to the investigational FMT, to ensure blinding during delivery.
  Other Names: FMP250; FMT
  Arms: Investigational FMT; Investigational FMT + psyllium fiber
Dietary Supplement: Psyllium Husk Powder — All subjects assigned to the fiber treatment arms will be required to take 1 teaspoon (approximately 5 grams) of psyllium husk powder twice a day (morning and night) for 8 weeks, beginning 3 days prior to Week 0 screening colonoscopy.
  Psyllium husk powder is the dried and powdered form of a psyllium seed coat.
  Arms: Investigational FMT + psyllium fiber; Placebo FMT +/- psyllium fiber

SUMMARY:
A double-blind, randomized, placebo-controlled clinical trial examining the efficacy and safety of Fecal Microbiota Transplantation (FMT) and high fiber supplementation in patients with active mild to moderate Ulcerative Colitis (UC). All enrolled subjects will provide serological, stool and mucosal specimen at each clinic visit to help further define the alterations in microbial profiles and immune cell function in response to psyllium fiber after FMT treatment.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled clinical trial with the following treatment assignments:

1. Investigational FMT (one-time)

   1. Subject will blindly receive investigational FMT once at day 0 colonoscopy
   2. Subjects in this group will blindly receive placebo FMP250 at week 8 by flexible sigmoidoscopy.
2. Investigational FMT (one-time) + Psyllium (2x/day for 8 weeks)

   1. Subject will blindly receive investigational FMT once at day 0 colonoscopy
   2. Subjects in this group will blindly receive placebo FMP250 at week 8 by flexible sigmoidoscopy.
3. Placebo FMT (one-time) +/- Psyllium (2x/day for 8 weeks)

   1. Subject will blindly receive placebo FMT once at day 0 colonoscopy
   2. Subjects in this group will blindly receive investigational FMP250 at week 8 by flexible sigmoidoscopy.

Subjects will blindly receive the investigational or placebo FMP250 treatment if they meet all inclusion and exclusion criteria during the day 0 screening colonoscopy. Subjects will receive follow-up phone calls at day 1, week 2, week 6, and week 10 post-FMT and will return for clinic visits at week 4, week 8 and week 12 post-FMT. Stool and blood samples will be collected for research purposes from subjects at every clinic visit (Day 0 colonoscopy, Week 4, Week 8, and Week 12). Mucosal biopsies will also be taken during the initial colonoscopy, at day 0 and during the follow-up flexible sigmoidoscopy at week 8. At week 8 post-FMT, all subjects will be evaluated by flexible sigmoidoscopy. Subjects originally randomized into the placebo cohort at week 0 will receive investigational FMP250 by flexible sigmoidoscopy at week 8, and subjects originally randomized into the investigational cohort at week 0 will receive placebo FMP250 by flexible sigmoidoscopy at week 8. Lastly, all subjects will be contacted for follow-up phone calls every subsequent 6 months for the next year.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female ≥ 18 years of age.
* Documentation of prior history of mild to moderate UC.
* Endoscopy confirmed active UC ≥ 15 centimeters at week 0 screening colonoscopy.

  a. As defined by a total Mayo scoring of 4-10 with an endoscopic sub-score ≥ 1.
* Patients must have a descending intact colon.
* Patients taking steroid or biologic therapy must be on a stable dose for 4 weeks prior to screening and maintained throughout the trial.
* Eligible patients willing to undergo screening testing prior to FMT to document baseline status:

  1. Urine Testing
  2. Blood Testing
  3. Stool Testing
* Patients must discontinue anti-rCDI antibiotics (e.g. vancomycin, fidaxomicin) 48 hours prior to FMT delivery procedure.

Exclusion Criteria:

* Biopsy proven Crohn's disease
* UC patients with severe disease (defined as a total mayo score >10)
* Clinical complications requiring emergent management (e.g. stricture, bowel obstruction, perforation and/or abscess)
* Concurrent C. difficile or other infections
* Primary sclerosing cholangitis
* Prior history of FMT
* Treatment for malignancy within past 5 years
* Active or latent tuberculosis
* Clinically meaningful laboratory abnormalities

  1. Hb: < 8
  2. ALT: greater than 3x the ULN (upper limit of normal)
* History of anaphylactic reactions to food allergens or allergy to psyllium husk
* Subject having any other condition that, in the opinion of the investigator, would jeopardize the safety or rights of the subject participating in the study, would make it unlikely for the subject to complete the study, or would confound the study.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2024-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randy Longman, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jacob V, Crawford C, Cohen-Mekelburg S, Viladomiu M, Putzel GG, Schneider Y, Chabouni F, O'Neil S, Bosworth B, Woo V, Ajami NJ, Petrosino JF, Gerardin Y, Kassam Z, Smith M, Iliev ID, Sonnenberg GF, Artis D, Scherl E, Longman RS. Single Delivery of High-Diversity Fecal Microbiota Preparation by Colonoscopy Is Safe and Effective in Increasing Microbial Diversity in Active Ulcerative Colitis. Inflamm Bowel Dis. 2017 Jun;23(6):903-911. doi: 10.1097/MIB.0000000000001132. PMID 28445246
- [Derived] Gogokhia L, Tran N, Grier A, Nagayama M, Xiang G, Funez-dePagnier G, Lavergne A, Ericsson C, Ben Maamar S, Zhang M, Battat R, Scherl E, Lukin DJ, Longman RS. Donor composition and fiber promote strain engraftment in a randomized controlled trial of fecal microbiota transplant for ulcerative colitis. Med. 2025 Sep 12;6(9):100707. doi: 10.1016/j.medj.2025.100707. Epub 2025 Jun 2. PMID 40460824

RESULTS

PARTICIPANT FLOW:
Groups:
- Investigational FMT: Participants will be blindly randomized to receive a single dose of investigational FMT during the week 0 colonoscopy.
  Additionally, participants will blindly receive a single dose of placebo FMT during the week 8 by flexible sigmoidoscopy.
  Fecal Microbiota Transplantation: The proposed intervention will deliver 250 milliliters of FMT by colonoscopy to the investigational FMT treatment groups at week 0. The placebo treatment group will instead receive the placebo FMT by colonoscopy at week 0 and then the investigational FMT by flexible sigmoidoscopy at week 8.
  Investigational FMT is biologically active human fecal material that is pre-screened, tested, quarantined, stored, packaged, and labeled by OpenBiome. Placebo FMP250 is a control unit made of glycerol, saline, and food dye that is stored, packaged, and labeled identically to the investigational FMT, to ensure blinding during delivery.
- Investigational FMT + Psyllium Fiber: Participants will be blindly randomized to receive a single dose of investigational FMT during the week 0 colonoscopy. They will also receive fiber supplementation of 1 teaspoon 2x/day for 8 weeks.
  Additionally, participants will blindly receive a single dose of placebo FMT during the week 8 by flexible sigmoidoscopy.
  Fecal Microbiota Transplantation: The proposed intervention will deliver 250 milliliters of FMT by colonoscopy to the investigational FMT treatment groups at week 0. The placebo treatment group will instead receive the placebo FMT by colonoscopy at week 0 and then the investigational FMT by flexible sigmoidoscopy at week 8.
  Investigational FMT is biologically active human fecal material that is pre-screened, tested, quarantined, stored, packaged, and labeled by OpenBiome. Placebo FMP250 is a control unit made of glycerol, saline, and food dye that is stored, packaged, and labeled identically to the investigational FMT, to ensure blinding during delivery.
  Psyllium Husk Powder: All subjects assigned to the fiber treatment arms will be required to take 1 teaspoon (approximately 5 grams) of psyllium husk powder twice a day (morning and night) for 8 weeks, beginning 3 days prior to Week 0 screening colonoscopy.
  Psyllium husk powder is the dried and powdered form of a psyllium seed coat.
- Placebo FMT +/- Psyllium Fiber: Participants will be blindly randomized to receive a single dose of placebo FMT during the week 0 colonoscopy. They may or may not also receive fiber supplementation of 1 teaspoon 2x/day for 8 weeks.
  Additionally, participants will blindly receive a single dose of investigational FMT during the week 8 by flexible sigmoidoscopy.
  Psyllium Husk Powder: All subjects assigned to the fiber treatment arms will be required to take 1 teaspoon (approximately 5 grams) of psyllium husk powder twice a day (morning and night) for 8 weeks, beginning 3 days prior to Week 0 screening colonoscopy.
  Psyllium husk powder is the dried and powdered form of a psyllium seed coat.
Period: Week 8 Colonoscopy
Arm/Group | Investigational FMT | Investigational FMT + Psyllium Fiber | Placebo FMT +/- Psyllium Fiber
Started | 9 | 9 | 9
Completed | 8 | 6 | 8
Not Completed | 1 | 3 | 1
Period: Follow Up
Arm/Group | Investigational FMT | Investigational FMT + Psyllium Fiber | Placebo FMT +/- Psyllium Fiber
Started | 9 | 9 | 9
Completed | 9 | 9 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Investigational FMT | Investigational FMT + Psyllium Fiber | Placebo FMT +/- Psyllium Fiber | Total
Number analyzed (Participants) | 9 | 9 | 9 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 8 | 25
  >=65 years | 0 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 8
  Male | 6 | 6 | 7 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 9 | 9 | 8 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 8 | 9 | 8 | 25
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 9 | 27

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response
Description: Clinical response at week 8 post-FMT, as defined by the reduction of the Mayo scoring system by >3 points (+30% reduction) with an accompanying decrease in the sub-score for rectal bleeding of at least 1 point
Time Frame: Week 8 post-FMT
Population: Analysis will be performed based on intent to treat. Therefore, any subjects with missing primary endpoint data at week 8 will have their baseline Mayo score carried forward to remain the same for the week 8 primary endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational FMT | Investigational FMT + Psyllium Fiber | Placebo FMT +/- Psyllium Fiber
Number analyzed (Participants) | 9 | 9 | 9
Participants | 5 | 2 | 1

2. Secondary Outcome: Clinical Remission
Description: Clinical remission at week 8 post-FMT, as defined by Mayo score ≤ 2 without any subscore >1
Time Frame: Week 8 post-FMT
Population: Analysis will be performed based on intent to treat. Therefore, any subjects with missing data at week 8 will have their baseline Mayo score carried forward to remain the same for the evaluation of clinical remission at week 8.
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational FMT | Investigational FMT + Psyllium Fiber | Placebo FMT +/- Psyllium Fiber
Number analyzed (Participants) | 9 | 9 | 9
Participants | 3 | 1 | 0

3. Secondary Outcome: Endoscopic Response or Remission
Description: Endoscopic response or remission at week 8 post-FMT, as defined by a Mayo endoscopic sub-score 0-1 with at least a 1-point reduction from baseline or a Mayo endoscopic sub-score of 0
Time Frame: Week 8 post-FMT
Population: Analysis will be performed based on intent to treat. Therefore, any subjects with missing data at week 8 will have their baseline Mayo score carried forward to remain the same for the evaluation of endoscopic response and remission at week 8.
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational FMT | Investigational FMT + Psyllium Fiber | Placebo FMT +/- Psyllium Fiber
Number analyzed (Participants) | 9 | 9 | 9
Participants | 4 | 2 | 0

4. Secondary Outcome: Number of Treatment or Disease Related Adverse Events.
Description: Adverse event counts are cumulative frequencies of adverse and severe adverse events assessed at Week 0 Colonoscopy - Week 12 post-FMT, 6 months post-FMT, and 1 year post-FMT.
Time Frame: Week 0 Colonoscopy - Week 12 post-FMT, 6 months post-FMT, and 1 year post-FMT
Measure: Number; unit: Adverse and Severe Adverse Events
Arm/Group | Investigational FMT | Investigational FMT + Psyllium Fiber | Placebo FMT +/- Psyllium Fiber
Number analyzed (Participants) | 9 | 9 | 9
Adverse and Severe Adverse Events | 21 | 33 | 20

ADVERSE EVENTS:
Time Frame: Adverse event data was collected up to 12 weeks post-FMT. Serious adverse event data was also collected at 6 months and 1 year.
Arm/Group | Investigational FMT | Investigational FMT + Psyllium Fiber | Placebo FMT +/- Psyllium Fiber
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 4/9 | 7/9 | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational FMT (N=9) | Investigational FMT + Psyllium Fiber (N=9) | Placebo FMT +/- Psyllium Fiber (N=9)
Worsening ulcerative colitis disease activity (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Investigational FMT (N=9) | Investigational FMT + Psyllium Fiber (N=9) | Placebo FMT +/- Psyllium Fiber (N=9)
Diarrhea (Gastrointestinal disorders) | 2 | 3 | 3
Abdominal Pain (Gastrointestinal disorders) | 2 | 3 | 2
Nausea (Gastrointestinal disorders) | 2 | 2 | 2
Fever (General disorders) | 1 | 3 | 2
Fatigue (General disorders) | 2 | 3 | 0
COVID-19 Infection (Infections and infestations) | 0 | 4 | 1
Chills (General disorders) | 2 | 0 | 2
Bloating (Gastrointestinal disorders) | 2 | 2 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1 | 2
Headache (General disorders) | 0 | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 2 | 0
Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Vomiting (General disorders) | 1 | 1 | 1
Yersinia Enterocolitis Infection (Infections and infestations) | 0 | 2 | 0
Fecal Urgency (Gastrointestinal disorders) | 1 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1
Stye Infection (Infections and infestations) | 0 | 0 | 1
Appetite Loss (General disorders) | 1 | 0 | 0
Hypotension (General disorders) | 1 | 0 | 0
Body Aches (General disorders) | 0 | 1 | 0
Enteropathogenic E. Coli Infection (Infections and infestations) | 0 | 1 | 0
Ear Infection (Infections and infestations) | 0 | 1 | 0
Eye Infection (Infections and infestations) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-11-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT03998488/Prot_SAP_002.pdf
  • Informed Consent Form (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT03998488/ICF_001.pdf